CLINICAL TRIAL: NCT06758167
Title: RCT Study on the Therapeutic Effect of Escitalopram Loaded With XingpiJieyu Formula on Resting State EEG Energy Abnormalities in Severe Liver Depression and Spleen Deficiency Type MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xueqin Wang, Principal Investigator, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-37-1
Record Dates: First submitted 2024-12-25; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Major Depression
Keywords: Depression; XingpiJieyu Formula; Escitalopram; Relative Energy; Electroencephalogram
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- XingpiJieyu formula (Experimental): Experimental group, treated with XingpiJieyu formula and escitalopram.
  Interventions: Drug: XingpiJieyu formula; Drug: Escitalopram
- Placebo and escitalopram (Placebo Comparator): Control group, treated with placebo and escitalopram.
  Interventions: Drug: Placebo; Drug: Escitalopram

INTERVENTIONS:
Drug: XingpiJieyu formula — XingpiJieyu formula is a traditional Chinese medicine. It pays attention to the regulation of qi and blood. Previous studies have shown that its clinical effect of treating mild and moderate depression is significant, for example, it can effectively improve depressive mood and somatic symptoms, and increase peripheral blood ATP levels in patients with depression.
  Other Names: XPJYF
  Arms: XingpiJieyu formula
Drug: Placebo — Placebo, no therapeutic effect.
  Other Names: PLA
  Arms: Placebo and escitalopram
Drug: Escitalopram — A commonly used drug in MDD treatment.
  Other Names: ESC

SUMMARY:
To compare the clinical efficacy of XingpiJieyu formula or its placebo combined with Escitalopram (ESC) in the treatment of moderate and severe MDD, and to explore a new method of integrated traditional Chinese and western medicine for the treatment of moderate and severe MDD with severe liver depression and spleen deficiency, as well as its neurological mechanism for regulating the relative power (RP) of resting-state EEG spectra.

DETAILED DESCRIPTION:
MDD patients, especially severe MDD patients have heavy burden of disease, high risk of suicide, difficulty in single drug treatment, and poor compliance with combined western medicine treatment. It is urgent to explore new methods of integrated traditional Chinese and western medicine in the treatment of moderate and severe MDD to enhance efficacy and reduce toxicity. A double-blind, randomized, controlled Trial (RCT) was conducted to compare the efficacy of XingpiJieyu formula or its placebo combined with escitalopram in the treatment of MDD with severe liver depression and spleen deficiency. We aim to explore the clinical efficacy of XingpiJieyu formula combined with escitalopram and its possible multi-target neural mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. outpatient/inpatient, age 18-45 years old, right-handed;
2. western medical diagnosis meets the diagnostic criteria of MDD in DSM-5, without psychiatric features;
3. In accordance with the diagnostic criteria of depression and liver-stagnation and spleen-deficiency in the "Guidelines for Diagnosis and Treatment of Internal Diseases in Traditional Chinese Medicine" issued by the China Association of Chinese Medicine in 2008;
4. 17-item Hamilton Depression Scale score ≥18;
5. educational experience ≥5 years;
6. The current episode has not used antidepressants, antipsychotics, mood stabilizers, or other medications that can act on the central nervous system for at least 4 weeks;
7. Have not received physical therapy, such as MECT, rTMS, etc., in the past 6 months;
8. The total duration of the disease ≤10 years.

Exclusion Criteria:

1. Any current or previous mental disorder other than MDD according to DSM-5;
2. Diagnosis of syndromes other than depression and liver-stagnation and spleen-deficiency in the "Guidelines for Diagnosis and Treatment of Internal Diseases in Traditional Chinese Medicine" issued by the China Association of Chinese Medicine in 2008;
3. Suicidal ideation or suicidal behaviour (HAMD-17 item 3 > 2);
4. Drinking alcohol in the week prior to the enrollment;
5. Patients with neurological disorders, somatic disorders, organic brain diseases, and tumour;
6. Sleep disorders other than insomnia disorders currently diagnosed according to DSM-5, such as obstructive sleep apnea syndrome, periodic limb movement disorder, restless legs syndrome, etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Scale (HAMD-17) | 8 weeks
  The Hamilton Depression Scale (HAMD) was developed by Hamilton in 1960 and is the most commonly used scale for clinical assessment of depressive states. This scale is used by two trained raters to conduct a combined HAMD examination of the patient, usually in the form of conversation and observation, and at the end of the examination, the two raters rate independently; by using this scale, the severity of the condition and the effectiveness of the treatment can be evaluated.
Hamilton Anxiety Scale (HAMA) | 8 weeks
  Hamilton Anxiety Scale (HAMA), compiled by Hamilton in 1959, is one of the commonly used scales in psychiatric clinics, and the total score of HAMA can better reflect the severity of anxiety symptoms, which can be used to evaluate the severity of anxiety symptoms in patients with anxiety and depression disorders and to assess the effects of various medications and psychological interventions.
Health Questionnaire-15 (PHQ-15) | 8 weeks
  The Patient Health Questionnaire-15 (PHQ-15) is a scale used to assess an individual's somatic symptoms and dysfunction. It consists of 15 common somatic symptom items, and assesses a person's somatic health status by asking the participant to select the symptoms that correspond to his or her condition. The scale can be used to screen and assess the presence and severity of clusters of somatic symptoms, helping healthcare professionals to quickly understand a patient's somatic health problems.
Pittsburgh sleep quality index (PSQI) | 8 weeks
  The Pittsburgh sleep quality index (PSQI) was compiled in 1989 by Dr Buysse, a psychiatrist at the University of Pittsburgh, USA, and others. The scale is suitable for patients with sleep disorders and patients with psychiatric disorders to evaluate the quality of sleep, but also for the general population to assess the quality of sleep.
Treatment Emergent Symptom Scale (TESS) | 8 weeks
  The Side Effects Scale (TESS) is a tool used to assess side effects of medications. It rates side effects in different categories to determine the extent to which a drug is causing side effects in a patient and whether adjustments to the treatment regimen are needed. It can help physicians better understand the side effects of medications and make timely adjustments to treatment regimens to improve outcomes and reduce adverse reactions in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqin Wang, Doctor, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No